CLINICAL TRIAL: NCT01299441
Title: Noninvasive ECOM Monitoring of Hemodynamic Parameters During Liver Transplantation
Brief Title: Endotracheal Cardiac Output Monitor (ECOM) for Patients Undergoing Liver Transplantation
Status: Terminated | Type: Observational
Why Stopped: unable to complete statistical analysis
Sponsor: Mayo Clinic (Other)
Collaborators: CONMED Corporation (Industry)
Responsible Party: Principal Investigator, Timothy S. Shine, M.D., PI, Mayo Clinic
Other Study IDs: 10-007600
Record Dates: First submitted 2011-02-09; First posted 2011-02-18 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- OLT patients intubated with ECOM ETT: Patients undergoing liver transplantation and intubated with ECOM endotracheal tube (ETT).
  Interventions: Device: ECOM ETT

INTERVENTIONS:
Device: ECOM ETT — Intubation with ECOM endotracheal tube (ETT)

SUMMARY:
The purpose of this study is to determine whether the endotracheal cardiac output monitor (ECOM) is accurate and predictive in liver failure patients with hyperdynamic circulatory changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing liver transplantation surgery

Exclusion Criteria:

* Patients who are anticipated to remain intubated postoperatively for greater than 24 hours.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver transplantation
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
endotracheal cardiac output monitor (ECOM), a non-invasive cardiac output monitor, is accurate and predictive | Less than 24 hours
  Pulmonary artery catheters are a standard of care for intraoperative hemodynamic assessment during liver transplantation. We propose to compare hemodynamic parameters obtained from PA catheters and ECOM. Use the endotracheal cardiac output monitor (ECOM) to evaluate multiple hemodynamic parameters (invasive blood pressure from the indwelling arterial catheter, noninvasive cardiac output via ECOM), and compare these to the parameters obtained from PA catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Shine, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States